CLINICAL TRIAL: NCT00629460
Title: A Pilot Study of PET-CT in the Assessment of Pulmonary Nodules in Children With Malignant Solid Tumors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PETPUL
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Nodules
Keywords: Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: there is only one group/cohort. This is a non-therapeutic study.

SUMMARY:
Because the management of children with solid tumors hinges on the extent of disease, it is crucial to identify metastatic sites. Helical chest computed tomography (CT) is the standard method of excluding pulmonary metastases. However, CT lacks molecular information regarding nodule histology and often biopsy is required to exclude malignancy. Biopsy procedures carry known risks including those associated with anesthesia and sedation, infection, pneumothorax, hemorrhage, pain and other post-procedure and post-operative complications and may also add unnecessary cost to the management of the patient. We found that the ability of three experienced pediatric radiologists to correctly predict nodule histology based on CT imaging features was limited (57% to 67% rate of correct classification). Also, there was only slight to moderate agreement in nodule classification between these reviewers.

Furthermore, of 50 children who have undergone pulmonary nodule biopsy at St. Jude in the last five years, 44% (22/50) had only benign nodules.

Adult studies have shown that a nuclear medicine scan called fluoro-deoxyglucose (FDG) positron emission tomography (PET) and the fusion modality PET-CT are superior to diagnostic CT in distinguishing benign from malignant pulmonary nodules because FDG PET gives information about the metabolic activity of the nodule. Nodules that are malignant have more metabolic activity, hence more FDG uptake/intensity, than those that are benign. There has been little work done in children to determine the value of PET or PET-CT in the evaluation of pulmonary nodules.

DETAILED DESCRIPTION:
In this study, we seek to assess the feasibility of performing PET-CT for the evaluation of pulmonary nodules in children to obtain preliminary data for sample size determination for a larger multi-institutional trial. The primary objective of the multi-institutional trial will be to compare the accuracy of diagnostic CT alone to PET-CT in distinguishing benign from malignant nodules in children with solid malignancies. We are hopeful that PET-CT will allow us to better direct the clinical management of these patients and to reduce the number of invasive procedures performed to confirm the presence of benign disease.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a known or clinically suspected solid malignancy (excluding brain tumor)
* Nodule must be discovered at the time of diagnosis of the primary malignancy or after the completion of therapy

Exclusion Criteria:

* Participant has not been off therapy for at least 3 weeks before undergoing PET-CT

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with known or suspected malignant solid tumors found by CT to have at least one pulmonary nodule measuring> or equal to 0.5 cm and < or equal to 3.0 cm in size will be eligible for enrollment.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of performing PET-CT for the evaluation of pulmonary nodules in children with solid malignancies and to obtain preliminary data for sample size determination for a larger, multi-institutional prospective study. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McCarville, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- Mary E. McCarville, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org